CLINICAL TRIAL: NCT02542410
Title: Dopamine Receptor Agonist Therapy for Pain Relief in Women Suffering From Endometriosis: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Amy DiVasta, MD, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00018628
Record Dates: First submitted 2015-08-11; First posted 2015-09-07 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Cabergoline; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Norethindrone acetate 5 mg po daily x 6 months
  Interventions: Drug: Norethindrone acetate
- Experimental (Experimental): cabergoline 0.5 mg PO twice weekly x 6 months
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline
  Other Names: Dostinex
  Arms: Experimental
Drug: Norethindrone acetate
  Other Names: Aygestin
  Arms: Control

SUMMARY:
The proposed pilot study will estimate the efficacy and safety of a novel therapeutic agent, cabergoline, with a clinical standard therapy, norethindrone acetate, for the treatment of endometriosis-associated pain in young women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Surgically confirmed endometriosis
* Age between 15-40 y, and premenopausal
* Pelvic pain score ≥3 on a Visual Analog Scaleover the last month

Exclusion Criteria:

* Use of other concurrent hormone medications (such as birth control pills)
* Impaired liver function (ALT > 2x normal) or liver disease (cirrhosis, hepatitis)
* Pregnancy
* Breast cancer
* Active thromboembolic disease
* Uncontrolled hypertension, history of cardiac valve disorder, history of fibrotic disorders

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] DiVasta AD, Stamoulis C, Gallagher JS, Laufer MR, Anchan R, Hornstein MD. Nonhormonal therapy for endometriosis: a randomized, placebo-controlled, pilot study of cabergoline versus norethindrone acetate. F S Rep. 2021 Jul 24;2(4):454-461. doi: 10.1016/j.xfre.2021.07.003. eCollection 2021 Dec. PMID 34934987

RESULTS

PARTICIPANT FLOW:
Groups:
- Norethindrone Acetate 5 mg Daily: Norethindrone acetate 5 mg po daily x 6 months
  Norethindrone acetate
- Cabergoline 0.5 mg Twice Weekly: cabergoline 0.5 mg PO twice weekly x 6 months
  Cabergoline
Period: Overall Study
Arm/Group | Norethindrone Acetate 5 mg Daily | Cabergoline 0.5 mg Twice Weekly
Started | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Norethindrone acetate 5 mg po daily x 6 months
  Norethindrone acetate
- Experimental: cabergoline 0.5 mg PO twice weekly x 6 months
  Cabergoline
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 25.2 (8.7) | 24.8 (2.8) | 24.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Score in Worst Pain Over the Last Month
Description: visual analog scale, minimum=0 and maximum=10 Higher numbers are a worse outcome
  Outcome measures is calculated as the value at 6 months minus value at baseline.
Time Frame: Baseline, 6 months
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Norethindrone Acetate 5 mg: Norethindrone acetate 5 mg po daily x 6 months
  Norethindrone acetate
- Cabergoline 0.5 mg: cabergoline 0.5 mg PO twice weekly x 6 months
  Cabergoline
Arm/Group | Norethindrone Acetate 5 mg | Cabergoline 0.5 mg
Number analyzed (Participants) | 4 | 5
score on a scale | -0.5 (1.5) | -5 (2.5)

2. Secondary Outcome: Changes in Pain Interference Scores
Description: Brief Pain Inventory Interference subscale is a 7-item self-report measure, designed to assess the extent to which pain interferes with various components of functioning, including physical and emotional functioning and sleep.The items in this scale can be grouped into those that assess physical functioning (general activity; walking ability; normal work, including both work outside the home and housework), those that assess emotional functioning (mood; relations with people; enjoyment of life), and a single item that assess the extent to which pain interferes with sleep. The arithmetic mean of the seven interference items is used as a measure of pain interference (i.e., how much a participant's pain interferes with her ability to complete activities of daily living and functioning). The score on the pain interference subscale ranges from 0-70. Higher scores are worse outcomes.
  Outcome measure calculated as the value at 6 months minus the value at baseline
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Norethindrone Acetate 5 mg | Cabergoline 0.5 mg
Number analyzed (Participants) | 4 | 5
units on a scale | 0.85 (1.1) | 0 (1.1)

ADVERSE EVENTS:
Time Frame: 6 MONTHS
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=4) | Experimental (N=5)
IRREGULAR VAGINAL BLEEDING (Reproductive system and breast disorders) | 2 (2) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 5 (5)
FATIGUE (General disorders) | 1 (1) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT02542410/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT02542410/SAP_001.pdf